CLINICAL TRIAL: NCT01183949
Title: A Phase I/II Open-label Multicenter Study of AT7519M Alone and in Combination With Bortezomib in Patients With Previously Treated Multiple Myeloma
Brief Title: Effect of AT7519M Alone and AT7519M Plus Bortezomib in Patients With Previously Treated Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Collaborators: Multiple Myeloma Research Consortium (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT7519M/0004
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma
Keywords: Neoplasms; Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Hemostatic Disorders; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases; Bortezomib; Antineoplastic Agents
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Hemostatic Disorders; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Patients will be enrolled into 3 groups which will run sequentially. Groups A and B will receive AT7519M only, whereas Group C will receive AT7519M in combination with Bortezomib.
  Interventions: Drug: AT7519M; Drug: Bortezomib

INTERVENTIONS:
Drug: AT7519M — Part A: Nine patients will receive AT7519M as an intravenous infusion on days 1, 4, 8 and 11 of a three week cycle. The starting dose of AT7519M will be 21mg/m^2/dose and will be increased to 27mg/m^2/dose during subsequent cycles in the absence of AT7519M-related toxicities.
  Part B: Amendment clarified there will be no further exploration of AT7519M as a monotherapy.
  Part C: Amendment modified dose escalation to a conventional 3 + 3 design with a maximum total of 14 patients will be treated at the maximum tolerated dose.
Drug: Bortezomib — Part C will treat between 3-26 patients with a combination of bortezomib and AT7519M in a dose escalation design. The starting doses for the dose escalation are bortezomib 1 mg/m2 and AT7519M 14 mg/m2.

SUMMARY:
The purpose of this study is to determine whether AT7519M alone or AT7519M plus bortezomib are effective treatments in patients with previously treated multiple myeloma.

DETAILED DESCRIPTION:
The clinical study AT7519M/0004 is an open-label multicenter study to investigate the efficacy of AT7519M alone and AT7519M in combination with bortezomib in patients with previously treated multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the risks of the study and provide signed informed consent
* Age 18 years or older
* Relapsed and or Refractory MM
* Disease progression following at least two systemic treatments for MM
* Patient must be refractory to the last bortezomib
* ECOG performance status 0, 1 or 2

Exclusion Criteria:

* Pregnant or lactating females. Patients of childbearing potential must use appropriate birth control throughout the study
* Inadequate liver function
* Renal impairment
* Neutrophil count <1.0 x 10^9 /litre in the absence of growth factors
* Platelet count <50 x 10^9 /litre in patients in whom <50% of bone marrow nucleated cells are plasma cells and <30 x 10^9 /litre in patients in whom ≥50 % of bone marrow nucleated cells are plasma cells
* Hemoglobin <8g/dl in the absence of transfusion
* Treated corrected calcium >ULN
* Serum creatine phosphokinase >ULN
* All previous cytotoxic therapies for MM must have been completed at least four weeks prior to treatment with AT7519M (two weeks for all non-cytotoxic therapy)
* Patients may be receiving concomitant therapy with biphosphonates and low dose corticosteroids. Bisphosphonates doses should be stable for at least 30 days prior to study drug administration. Corticosteroids doses should be stable for at least 7 days prior to study treatment
* Prior peripheral stem cell transplant within 12 weeks
* Evidence of mucosal or internal bleeding and/or platelet transfusion refractory (unable to maintain a platelet count >50 x 10^9 /litre)
* Ongoing infection requiring treatment
* Previous radiotherapy within 2 weeks of the start of the study
* Having previously received treatment with a cyclin-dependent kinase or GSK3beta inhibitor
* Incomplete recovery from previous radiotherapy other than residual cutaneous effects or stable < Grade 2 gastrointestinal toxicity
* Prior radiotherapy to the head and neck region for head and neck tumors
* Previous malignancy, except for non-melanomatous skin carcinomas, in situ carcinomas or malignancies with low risk of recurrence.
* Any severe or uncontrolled systemic conditions (e.g. systemic infection) or current unstable or uncompensated respiratory or cardiac conditions which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol
* Incomplete recovery from surgery other than stable < Grade 2 toxicity
* Peripheral neuropathy > Grade 2
* Abnormal left ventricular ejection fraction (< lower limit of normal for the institution for a patient of that age) on echocardiogram
* History of an ischemic cardiac event, including myocardial infarction within 3 months of study entry
* Congestive cardiac failure of ≥ grade 3 severity according to NYHA functional classification
* Unstable cardiac disease
* History or presence of bradycardia (≤60bpm), left bundle branch block, heart block, cardiac pacemaker or significant atrial tachyarrhythmias
* If the patient will receive bortezomib (Velcade) during part C of the study, concurrent treatment with any medication known strongly to inhibit or induce CYP3A4, CYP1A2 and CYP2C19 which cannot be discontinued at least two week prior to treatment with AT7519M (other than corticosteroids)
* Concurrent treatment with any medication that prolongs QT interval and may induce Torsades de Pointes and which cannot be discontinued at least two weeks prior to treatment with AT7519M
* Family or personal history of long QTc syndrome or ventricular arrhythmias including ventricular bigeminy
* Previous history of drug-induced QTc prolongation
* Screening 12-lead ECG with measurable QTc interval according to Fridericia's Correction of >450 msecs
* Screening 12-lead ECG with ST depression >1 mm in 2 or more leads or T wave inversion in 2 or more contiguous leads
* Prior history of infection with human immunodeficiency virus (HIV), known active hepatitis B or C viruses
* Diffuse infiltrative pulmonary or pericardial disease
* Known hypersensitivity to bortezomib, boron or any of the excipients of VelcadeTM
* Epilepsy or other convulsive disorder requiring active management
* Serious psychiatric illness, active alcoholism or drug addiction that may hinder or confuse follow up evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-11; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical efficacy of AT7519M alone or in combination with bortezomib | Subjects with be followed until disease progression (an average of 4 cycles per subject. i.e an average of 84 days)
  Efficacy will be assessed using the International Multiple Myeloma Working Group (IMWG) Response Criteria

SECONDARY OUTCOMES:
Assess the type, incidence and severity of clinically significant treatment emergent adverse events as assessed by National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) V 4.03 | Subjects with be followed until disease progression (an average of 4 cycles per subject, i.e an average of approximately 84 days)
To define the pharmacokinetic profile of AT7519M and bortezomib when administered alone or in combination with bortezomib | 2 cycles (i.e an average of 42 days)
  The pharmacokinetic evaluation will include the calculation of plasma clearance and elimination phase half-life for AT7519M and bortezomib
To identify the maximum tolerated dose (MTD) of AT7519M in combination with bortezomib | Subjects with be followed until disease progression (an average of 4 cycles per subject, i.e an average of approximately 84 days)
  The MTD will be based on the incidence of dose limiting toxicities

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Faber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Centre, New York, New York
  - MCW and Froedtert Clinical Cancer Center, Division of Neoplastic Diseases & Related Disorders, Milwaukee, Wisconsin